CLINICAL TRIAL: NCT00933920
Title: A Randomized, Single-blind, Parallel Group, Multiple Oral Dose Study to Evaluate the Effect of a Light Meal on the Pharmacokinetics and Pharmacodynamics of Aliskiren Using Market 300 mg Tablet Formulation in Subjects With Mild to Moderate Hypertension
Brief Title: Effect of Light Meal on Pharmacokinetic and Pharmacodynamics of Aliskiren in Patients With Mild to Moderate Hypertension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: CSPP100A2110; CTRI/2009/091/000287; 26-06-2009
Record Dates: First submitted 2009-07-03; First posted 2009-07-07 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2010-02

CONDITIONS: Hypertension
Keywords: Aliskiren,; hypertension,; renin-angiotensin-aldosterone system,; pharmacokinetics,; pharmacodynamics
MeSH Terms: conditions — Hypertension | interventions — aliskiren

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Fed Group (Active Comparator)
  Interventions: Drug: Aliskiren
- Fasted group (Active Comparator)
  Interventions: Drug: Aliskiren

INTERVENTIONS:
Drug: Aliskiren
  Arms: Fed Group
Drug: Aliskiren
  Arms: Fasted group

SUMMARY:
The purpose of this study is to determine the effect of a light meal on the pharmacokinetics and pharmacodynamics of aliskiren in patients with mild to moderate hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients, 18 to 65 years of age with mild to moderate hypertension
* Patients who are eligible and able to participate in the study

Exclusion criteria:

* Severe hypertension
* Secondary form of hypertension.
* Type 1 or type 2 diabetes mellitus
* Serum potassium out side laboratory reference range
* Any history of hypertensive encephalopathy or cerebrovascular accident

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2009-06; Primary Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Compare PK (AUC & Cmax) and PD, i.e. PRA (Plasma Renin Activity, AUE) of aliskiren when given with and without light meal. | 28 Days

SECONDARY OUTCOMES:
Compare the effect of Plasma Renin Concentration (PRC) and angiotensin II of aliskiren when given with and without light meal | 28 Days
Assess safety and tolerability of aliskiren when given with and without light meal | 28 days
Evaluate the effect on mean sitting systolic and diastolic blood pressure of aliskiren when given with or without a light meal | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- India (5):
  - Novartis Investigator Site, Coimbatore
  - Novartis Investigative Site, Hyderabaad
  - Novartis Investigator Site, Hyderabaad
  - Novartis Investigator Site, Mangalore
  - Novartis Investigative Site, New Delhi

REFERENCES:
- See also: Results for CSPP100A2110 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=3763